CLINICAL TRIAL: NCT01519947
Title: Comparative Study to Evaluate the Effect of the Altitude on Dosage Requirements of Methoxy Polyethylene Glycol-Epoetin Beta to Correct Hemoglobin Levels in Chronic Renal Anemia in Pre-Dialysis and Dialysis Patients
Brief Title: A Study of The Effect of Altitude on Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) Dose Requirements in Participants With Chronic Renal Anemia in Pre-Dialysis or Dialysis
Acronym: ALTITUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25754
Record Dates: First submitted 2012-01-18; First posted 2012-01-27 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Anemia, Kidney Disease, Chronic
MeSH Terms: conditions — Anemia; Kidney Diseases; Bronchiolitis Obliterans Syndrome | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-dialysis, sea level (Active Comparator): Participants received 50-250 mcg SC according to local label.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta
- Dialysis, sea level (Active Comparator): Participants received 50-250 mcg SC according to local label.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta
- Pre-dialysis, >1800 meters (Experimental): Participants received 50-250 mcg SC according to local label.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta
- Dialysis, >1800 meters (Experimental): Participants received 50-250 mcg SC according to local label.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Participants received 50-250 mcg SC according to local label
  Other Names: Mircera

SUMMARY:
This comparative, open-label, multicenter, parallel-group study evaluated the effect of altitude on the dose requirements of Mircera (methoxy polyethylene glycol-epoetin beta) to achieve a target hemoglobin concentration of 11-12 grams per deciliter (g/dL) in participants with chronic renal anemia in pre-dialysis and dialysis. Four groups of participants, at sea level (below 50 meters) or an altitude above 1800 meters, and pre-dialysis or dialysis, received 50-250 micrograms (mcg) Mircera subcutaneously (SC), according to the local prescribing label.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Chronic kidney disease stage III-IV or V
* Probable start of dialysis within 18 months (pre-dialysis group)
* Hemodialysis or peritoneal dialysis in a stable regimen for at least 3 months (dialysis group)
* Adequate iron status
* Females of childbearing potential must agree to use two effective methods of contraception during the study and for at least 2 months following the last dose of study drug

Exclusion Criteria:

* Failing renal allograft in place
* Acute or chronic bleeding within 8 weeks prior to screening
* Transfusion of red blood cells within 8 weeks prior to screening
* Poorly controlled hypertension, defined as hypertension that needs hospitalization to obtain control
* History of seizures, hemoglobinopathies and/or severe liver disease
* Active malignant disease, except for non-melanoma skin cancer
* Immunosuppressive therapy in the 12 weeks prior to screening
* Treatment with any other investigational agent or participation in a clinical trial within 28 days prior to enrolment
* Known hypersensitivity to Mircera (methoxy polyethylene glycol-epoetin beta) or any of its excipients
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Mexico (7):
  - Clínica San Cosme Centro Especializado en el Tratamiento de Enfermedades Renales S.C, Aguascalientes
  - Nefros Investigación S.C., Delegación Coyoacan
  - Centro de hemodialisis del norte S.C., Mexicali
  - Hospital Angeles Lindavista;Nefrologia, Mexico City
  - Hospital Star Medica Morelia, Morelia
  - Unidad De Dialisis La Loma S.C., Pureto Vallarta
  - Hospital Regional De Alta Especialidad De Veracruz; Nephrology, Veracruz

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 87 participants were enrolled in the study. One participant did not receive study drug.
Groups:
- Pre-dialysis, Sea Level: Participants received 50-250 mcg subcutaneously (SC) according to local label.
Period: Overall Study
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Started | 19 | 11 | 15 | 42
Completed | 17 | 7 | 8 | 34
Not Completed | 2 | 4 | 7 | 8
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2 | 1
Not completed — Peritoneal Dialysis Needed | 0 | 1 | 0 | 0
Not completed — Development of Anemia | 0 | 1 | 0 | 1
Not completed — Blood Transfusion | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2
Not completed — Poor Response | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters | Total
Number analyzed (Participants) | 19 | 10 | 15 | 42 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (15.1) | 38.5 (18.8) | 61.7 (15.6) | 56.5 (17.4) | 56.2 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 8 | 23 | 48
  Male | 8 | 4 | 7 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Dose Required to Achieve Target Hemoglobin of 11-12 g/dL
Time Frame: Up to approximately 20 months
Population: The intent-to treat (ITT) population included all enrolled participants who received at least one dose of study drug and had baseline and post-baseline measurements of the primary outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms (mcg)
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Number analyzed (Participants) | 19 | 10 | 15 | 42
micrograms (mcg) | 150.3 (69.0) | 194.7 (214.2) | 98.7 (22.5) | 66.6 (33.6)

2. Secondary Outcome: Change in Hemoglobin Concentration
Time Frame: From baseline to 6 months
Population: The intent-to treat (ITT) population included all enrolled participants who received at least one dose of study drug and had baseline and post-baseline measurements of the primary outcome measure. Data are reported for evaluable participants.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Number analyzed (Participants) | 19 | 3 | 8 | 34
grams per deciliter (g/dL) | 1.4 (0.8) | 2.5 (1.5) | 2.0 (0.8) | 2.4 (1.4)

3. Secondary Outcome: Percentage of Participants Achieving Target Hemoglobin Concentration 11-12 g/dL After 3 and 6 Months of Treatment
Time Frame: 3 and 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Number analyzed (Participants) | 19 | 10 | 15 | 42
percentage of participants
  3 months | 36.8 | 10.0 | 0.0 | 28.6
  6 months | 52.6 | 0.0 | 13.3 | 19.0

4. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug.
Time Frame: Up to approximately 20 months
Population: The safety population included all enrolled participants who received at least one dose of study drug and had a subsequent safety evaluation dose.
Measure: Number; unit: percentage of participants
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Number analyzed (Participants) | 19 | 10 | 15 | 42
percentage of participants | 84.2 | 90.0 | 66.7 | 85.7

5. Secondary Outcome: Percentage of Participants Requiring Dose Adjustments
Description: This outcome measure was not assessed.
Time Frame: Up to approximately 20 months
Population: Data were not collected.
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Incidence of Red Blood Cell Transfusions
Description: This outcome measure was not assessed.
Time Frame: Up to approximately 20 months
Population: Data were not collected.
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 20 months
Arm/Group | Pre-dialysis, Sea Level | Dialysis, Sea Level | Pre-dialysis, >1800 Meters | Dialysis, >1800 Meters
Serious Adverse Events (participants affected / at risk) | 1/19 | 3/10 | 2/15 | 6/42
Other Adverse Events (participants affected / at risk) | 16/19 | 9/10 | 10/15 | 36/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-dialysis, Sea Level (N=19) | Dialysis, Sea Level (N=10) | Pre-dialysis, >1800 Meters (N=15) | Dialysis, >1800 Meters (N=42)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Collapse cardiovascular (General disorders) | 0 | 0 | 0 | 1
Malignant neoplasm of ampulla of Vater (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Infusion site infection (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cerebral thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-dialysis, Sea Level (N=19) | Dialysis, Sea Level (N=10) | Pre-dialysis, >1800 Meters (N=15) | Dialysis, >1800 Meters (N=42)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Cardiac disorders) | 1 | 1 | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Endocrine disorders) | 0 | 1 | 0 | 4
Hypoglycaemia (Endocrine disorders) | 1 | 0 | 3 | 1
Diabetic retinopathy (Endocrine disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 2 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Peritonitis (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 3 | 8
Catheter related infection (General disorders) | 0 | 1 | 0 | 2
Face oedema (General disorders) | 1 | 0 | 2 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 7
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infusion site infection (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 1 | 0 | 7
Transferrin saturation decreased (Investigations) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood iron decreased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Oedema peripheral (Metabolism and nutrition disorders) | 7 | 2 | 4 | 8
Oedema (Metabolism and nutrition disorders) | 0 | 0 | 1 | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Generalised oedema (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 4
Vertigo (Nervous system disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Somnolence (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Lipoma of breast (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 2
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Pharyngotonsillitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pallor (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Eye operation (Surgical and medical procedures) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 6 | 4 | 2 | 19
Ecchymosis (Vascular disorders) | 0 | 1 | 0 | 3
Hypertensive crisis (Vascular disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.